CLINICAL TRIAL: NCT06761014
Title: Comparative Effects of Instrumental Assisted Soft Tissue Mobilization and Sustained Stretching on Pain, Range of Motion and Function Among Hockey Players With Quadratus Lumborum Tightness.
Brief Title: Comparative Effects of Instrumental Assisted Soft Tissue Mobilization and Sustained Stretching Among Hockey Players
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/24/0431
Record Dates: First submitted 2025-01-01; First posted 2025-01-07 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Sports Physical Therapy
Keywords: Quadratus lumborum muscle; Low back pain; IASTM; instrument-assisted soft tissue mobilization; Range of motion; Sustained stretching
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Intervention Model Description: Randomized Control design
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: Instrumental assisted soft tissue mobilization (Experimental): 11 participates will receive IASTM treatment for total of 40 more seconds.
  Interventions: Other: Instrumental assisted soft tissue mobilization
- Group B: Sustained stretching (Experimental): 11 participates will receive total of thirty seconds, divided into three sets of stretches at each intervention, with ten seconds of rest in between.
  Interventions: Other: Sustained stretching

INTERVENTIONS:
Other: Instrumental assisted soft tissue mobilization — instrument will be held at 45° angle and the IASTM treatment will be administered for about 20 seconds in a direction parallel to the muscle fibers being treated with deep strokes
  Arms: Group A: Instrumental assisted soft tissue mobilization
Other: Sustained stretching — The therapist will apply the pressure or ask to maintain the stretch. A total of thirty seconds, divided into three sets of stretches at each intervention, with ten seconds of rest in between
  Arms: Group B: Sustained stretching

SUMMARY:
Effect of instrumental assisted soft tissue mobilization over sustained stretching in hockey players on improving quadratus lumborum flexibility.

DETAILED DESCRIPTION:
To find the effect of instrumental assisted soft tissue mobilization over sustained stretching in hockey players on improving quadratus lumborum flexibility.

ELIGIBILITY:
Inclusion Criteria:

Age group of 16-26 years. Male and female Deficit of thoracolumbar Range of Motion with QL tightness Participates with moderate pain as per the ODI (20%-40%)

Exclusion Criteria:

Not fit in the age group Who have muscles injury from last 6 months Who have ODI score less than 20% Who do not involve QL tightness

Ages: 16 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 22 (Actual)
Dates: Start 2024-04-24 (Actual); Primary Completion 2025-01-10 (Estimated); Study Completion 2025-01-20 (Estimated)

PRIMARY OUTCOMES:
Oswestry Disability Index Questionnaire: | 4 weeks
  The Oswestry disability index (ODI), which is frequently used to evaluate reported limitations in individuals with low back pain, was employed to measure the disability index. It has two items about pain and eight items about activities of daily life. Each item has a point value between 0 and 5. The disability index increases with the overall score, which is represented as a percentage. A revised scale with nine items was utilized since it was determined that the sex life-related questions on the tenth item were inappropriate for persons of Korean descent. This test's test-retest reliability was ICC=0.85-0.94, and its intra-rater reliability was ICC=0.81-0.90.
NPRS | 4 weeks
  The score for each item ranges from 0 to 10, measured in units of length up to the location where the patient indicated the level of pain. NPRS is known to have a high sensitivity to pain and is proportional to the pain. This is the most widely used measurement method for chronic pain as well as acute pain with a good reliability.
Inclinometer: | 4 weeks
  Inclinometers are a commonly used instrument in clinical practice. The recordings from digital inclinometers could be more objective. Given its non-invasive nature, ease of use, and utility in evaluating lumbar or thoracolumbar range of motion. Inter-rater: ICC = 0.60, test-retest: r = 0.13-0.87.

CONTACTS AND LOCATIONS:
Overall Officials: Dania Zaheer, DPT, Principal Investigator — Riphah International University
Locations (1):
- Pakistan sports board, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Knezevic NN, Candido KD, Vlaeyen JWS, Van Zundert J, Cohen SP. Low back pain. Lancet. 2021 Jul 3;398(10294):78-92. doi: 10.1016/S0140-6736(21)00733-9. Epub 2021 Jun 8. PMID 34115979
- [Background] Barboza SD, Joseph C, Nauta J, van Mechelen W, Verhagen E. Injuries in Field Hockey Players: A Systematic Review. Sports Med. 2018 Apr;48(4):849-866. doi: 10.1007/s40279-017-0839-3. PMID 29299879
- [Background] Kim YK, Cho SY, Lee KH. Effects of transcutaneous electrical nerve stimulation and instrument-assisted soft tissue mobilization combined treatment on chronic low back pain: A randomized controlled trial. J Back Musculoskelet Rehabil. 2021;34(5):895-902. doi: 10.3233/BMR-200369. PMID 34092603
- [Background] Lee JH, Lee DK, Oh JS. The effect of Graston technique on the pain and range of motion in patients with chronic low back pain. J Phys Ther Sci. 2016 Jun;28(6):1852-5. doi: 10.1589/jpts.28.1852. Epub 2016 Jun 28. PMID 27390432
- [Background] Nazary-Moghadam S, Yahya-Zadeh A, Zare MA, Ali Mohammadi M, Marouzi P, Zeinalzadeh A. Comparison of utilizing modified hold-relax, muscle energy technique, and instrument-assisted soft tissue mobilization on hamstring muscle length in healthy athletes: Randomized controlled trial. J Bodyw Mov Ther. 2023 Jul;35:151-157. doi: 10.1016/j.jbmt.2023.04.079. Epub 2023 Apr 21. PMID 37330762
- [Background] Osailan A, Jamaan A, Talha K, Alhndi M. Instrument assisted soft tissue mobilization (IASTM) versus stretching: A comparison in effectiveness on hip active range of motion, muscle torque and power in people with hamstring tightness. J Bodyw Mov Ther. 2021 Jul;27:200-206. doi: 10.1016/j.jbmt.2021.03.001. Epub 2021 Mar 11. PMID 34391234
- [Background] El-Hafez HM, Hamdy HA, Takla MK, Ahmed SEB, Genedy AF, Abd El-Azeim ASS. Instrument-assisted soft tissue mobilisation versus stripping massage for upper trapezius myofascial trigger points. J Taibah Univ Med Sci. 2020 Mar 6;15(2):87-93. doi: 10.1016/j.jtumed.2020.01.006. eCollection 2020 Apr. PMID 32368203
- [Background] Gunn LJ, Stewart JC, Morgan B, Metts ST, Magnuson JM, Iglowski NJ, Fritz SL, Arnot C. Instrument-assisted soft tissue mobilization and proprioceptive neuromuscular facilitation techniques improve hamstring flexibility better than static stretching alone: a randomized clinical trial. J Man Manip Ther. 2019 Feb;27(1):15-23. doi: 10.1080/10669817.2018.1475693. Epub 2018 Aug 1. PMID 30692839